CLINICAL TRIAL: NCT02236897
Title: Metabotropic Glutamate Receptor 5 (mGluR5) Imaging in Amyotrophic Lateral Sclerosis (ALS) Patients and Healthy Volunteers
Brief Title: PET Imaging in ALS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: ALS Association (Other)
Responsible Party: Principal Investigator, Lyle W. Ostrow, MD, PhD, Assistant Professor of Neurology, Johns Hopkins University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NA_00073452
Record Dates: First submitted 2014-09-08; First posted 2014-09-11 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PET Scanning (Experimental): Imaging of mGluR5 using PET scanning
  Interventions: Other: PET Scanning

INTERVENTIONS:
Other: PET Scanning

SUMMARY:
This is a pilot study to evaluate a potential imaging biomarker for aiding diagnosis and monitoring progression of ALS, based on a well established basic science pathway, published human autopsy data, preliminary data in ALS mutant mice, and our recently published data using brain PET scans to image the metabotropic glutamate receptor type 5 (mGluR5) in healthy human volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ALS patients, ranging in age from 18-80.
* Must meet El Escorial Criteria for Probable or Definite ALS.
* Disease duration >1 year, but <3 years.
* Weakness in at least two extremities.
* Forced vital capacity less than 80% and greater than 50%.

Exclusion Criteria:

* Documented orthopnea or otherwise unable to lie flat in a PET scanner for 90 minutes.
* Presence of pacemakers, aneurysm clips, shrapnel, or other implanted metallic devices that would preclude an MRI scan.
* Absence of sufficient collateral arterial circulation for radial arterial line placement in both wrists.
* Significant abnormalities of hepatic or renal function, or illicit substance use.
* Positive drug screen. (Subjects currently taking prescribed narcotic medication who have a positive drug screen for this medication will not be excluded. Medication history will be obtained during screening).
* Weighs > 350 lbs.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-08; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Glutamate Receptor Distribution | 1 year
  The two primary outcome variables (VT and BPND) are quantitative estimates of mGluR5 distribution in the defined central nervous system regions. We will employ plasma reference graphical analysis (PRGA) which yielded the most accurate estimates of BPND and VT in a test-retest scheme. We will perform various analyses to determine if BPND or VT measurements in the volumes of interest differ between the ALS and control subject groups.

CONTACTS AND LOCATIONS:
Overall Officials: Lyle Ostrow, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States